CLINICAL TRIAL: NCT00001487
Title: Dehydroepiandrosterone Treatment of Mid-Life-Related Mood Disorders in Women and Men
Brief Title: Treatment of Mid-Life-Related Mood Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950151; 95-M-0151
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-04

CONDITIONS: Depressive Disorder; Mood Disorder
Keywords: Menopause; Andropause; Depression; DHEA; Steroids; Mid-Life Depression; Mid Life; Perimenopause; Climecteric-Related Mood Disorder
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depression | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: Dehydroepiandrosterone

SUMMARY:
Dehydroepiandrosterone (DHEA) is a hormone produced by the adrenal gland. As humans grow older the levels of DHEA naturally decrease. Low levels of DHEA have been associated with a variety of harmful effects, including increased heart disease, decreased immune system function, decreased bone density (osteoporosis), high cholesterol, and increased fat to muscle ratio.

Blood levels of DHEA and its sulfate form, DHEA-S, begin dropping when humans are in their 20's. By the time humans are in their 40's and 50's, levels of DHEA and DHEA-S levels are at 50% of their peak. Previous studies have shown that levels of these hormones are associated with feelings of "well-being" and enjoyment of "leisure" activities.

In this study researchers are interested in the effects on mood and behavior of DHEA in men and women with mid-life related mood disorders. Specifically, researchers would like to find out if increasing levels of DHEA will lessen the symptoms associated with these disorders.

DETAILED DESCRIPTION:
Dehydroepiandrosterone (DHEA) is a hormone produced by the adrenal gland in concentrations that decrease with age. In humans low DHEA levels have been associated with a variety of adverse biological consequences, including increased cardiovascular disease, decreased immune function, decreased bone density, negative lipid profile and an increased fat to muscle ratio.

In this study, we investigate the effects on mood and behavior of DHEA in men and women with midlife-related mood disorders in a double-blind, placebo-controlled, crossover trial. We specifically ask whether increasing DHEA levels will mitigate any or all of the neurasthenia-like symptoms characteristic of these disorders.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects for this study will meet the following criteria:

A current episode of minor (meeting 3-4 criterion symptoms) or major depression of moderate severity or less on the SCID severity scale for depression and not meeting DSM-IV criteria symptom #9 (suicide) as determined by the administration of the minor depression module of the SADS-L and the Structured Clinical Interview for DSM-IV. Additionally, to ensure that subjects meet a minimum threshold for severity of depression, subjects will have scores greater than or equal to 10 on either the Beck Depression Inventory (BDI) or the Center for Epidemiologic Studies - Depression (CES-D) Scale during at least three of the four clinic visits during the two month screening phase. Subjects will be excluded if they meet any of the following criteria: major depression of greater than moderate severity, DSM-IV criteria #9 (suicide), or anyone requiring immediate treatment after clinical assessment, functional impairment ratings of five or six for more than seven consecutive days on daily ratings;

Age 40-65;

No prior hormonal therapy for the treatment of menopause/andropause-related mood or physical symptoms within the last six months;

In good medical health.

EXCLUSION CRITERIA:

The following conditions will constitute contradictions to treatment with DHEA and will preclude a subject's participation in this protocol:

Positive (threshold) response to SCID major depression section item #9, suicidal ideation;

Anyone requiring immediate treatment after clinical assessment;

Severity ratings greater than moderate on the SCID;

Functional impairment ratings of five or six for more than seven consecutive days on daily ratings

Current treatment with antidepressant medications

Prostate nodules or cancer

Moderate symptoms of benign prostatic hypertrophy such as hesitancy, urgency, frequent voiding and feeling of incomplete voiding

History of ischemic cardiac disease

Renal disease

Hepatic dysfunction

Women with a history of carcinoma of the breast, or any women with a family history of the following: premenopausal breast cancer or bilateral breast cancer in a first degree relative; multiple family members (greater than three relatives) with postmenopausal breast cancer

Women with a history of uterine cancer

Patients with a known hypersensitivity to DHEA or other androgens

Pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-06; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bloch M, Schmidt PJ, Danaceau MA, Adams LF, Rubinow DR. Dehydroepiandrosterone treatment of midlife dysthymia. Biol Psychiatry. 1999 Jun 15;45(12):1533-41. doi: 10.1016/s0006-3223(99)00066-9. PMID 10376113
- [Background] Morales AJ, Nolan JJ, Nelson JC, Yen SS. Effects of replacement dose of dehydroepiandrosterone in men and women of advancing age. J Clin Endocrinol Metab. 1994 Jun;78(6):1360-7. doi: 10.1210/jcem.78.6.7515387.
- [Background] Schmidt PJ, Nieman L, Danaceau MA, Tobin MB, Roca CA, Murphy JH, Rubinow DR. Estrogen replacement in perimenopause-related depression: a preliminary report. Am J Obstet Gynecol. 2000 Aug;183(2):414-20. doi: 10.1067/mob.2000.106004. PMID 10942479